CLINICAL TRIAL: NCT01851499
Title: Ultramicronized PEA (Normast) in Spinal Cord Injury Neuropathic Pain: a Randomized, Double-blind, Placebo-controlled, Parallel, Multi-center Study
Brief Title: Ultramicronized PEA (Normast) in Spinal Cord Injury Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Pain Research Center (Other)
Collaborators: Spinal Cord Injury Centre of Western Denmark (Other); Glostrup University Hospital, Copenhagen (Other); Epitech Group SRL, Italy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Normast-2013
Record Dates: First submitted 2013-05-08; First posted 2013-05-10 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Neuropathic Pain; Spinal Cord Injury
Keywords: Neuropathic pain following spinal cord injury
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultramicronized PEA (Normast) (Experimental): Normast is ultramicronized Palmitoylethanolamide (PEA) classified as "Dietary foods for special medical purposes".
  Interventions: Dietary Supplement: Ultramicronized PEA (Normast)
- Microgranules (Placebo Comparator): Same as Normast, without active component.
  Interventions: Dietary Supplement: Ultramicronized PEA (Normast)

INTERVENTIONS:
Dietary Supplement: Ultramicronized PEA (Normast) — 600 mg

SUMMARY:
Randomized, double-blinded, placebo-controlled, parallel group study of ultramicronized PEA (Normast)600 mg x 2 daily or corresponding placebo with a week of baseline period followed by 1 x 12 weeks treatment period.

DETAILED DESCRIPTION:
Study design: Randomized, double-blinded, placebo-controlled, parallel, multi-center study of ultramicronized PEA (Normast)with a week of baseline period followed by 1 x 12 weeks treatment period.

Methodology: Given Normast 600mg x 2 daily or corresponding placebo and kept on that dose for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or more with at- and/or below-level neuropathic pain for at least 3 months due to trauma or disease of the spinal cord or cauda equina (of at least 6 months old) with a mean pain intensity from 4 to 9 on a 0-10 point numeric rating scale (NRS) during a one-week baseline period will be eligible for the study

Exclusion Criteria:

* known concomitant severe cerebral damage, terminal illness, planned surgery, pregnancy or lactation, alcohol or substance abuse, hypersensitivity to PEA or carrier, and psychiatric disease except depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2013-05; Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in mean pain intensity on a 0-10 numerical rating scale from baseline week to last week of treatment | 12 weeks

SECONDARY OUTCOMES:
Spasticity/spasms and sleep disturbance, change in mean score from baseline to last week of treatment | 12 weeks
Modified Tardieu and clonus over ankle joints | 12 weeks
Spasticity and spasms on a 0-10 NRS | 12 weeks
Health related quality of life S-TOPS | 12 weeks
Global Impression of Change | 12 weeks
Pain relief of overall pain and at-and below level pain | 12 weeks
allodynia(touch and cold) | 12 weeks
Pain symptoms evaluated by NPSI | 12 weeks
pain impact on activities, sleep and mood | 12 weeks
effect on unpleasantness | 12 weeks
escape medication | 12 weeks
Insomnia Severity Index | 12 weeks
anxiety(GAD-10) | 12 weeks
depression(MDI) | 12 weeks
NNT for 33% and 50% pain reduction | 12 weeks
Combined spasticity and pain score (CPSS) | 12 weeks
Numbers of responders (33% pain reduction) in those with and without allodynia/hyperalgesia and those with different pain symptoms (NPSI) | 12 weeks

OTHER OUTCOMES:
Blindness is assessed by asking the patients and treating physician which treatment they believed they recieved and the reason for this | 12 weeks
Number of patients with adverse events and number, type and severity of adverse events. | 12 weeks
  Adverse events are assessed using open-ended questions both during and after treatment period.
  SAE reporting will be performed according to GCP and regulatory requirements.

CONTACTS AND LOCATIONS:
Overall Officials: Sven R. Andresen, MD, Principal Investigator — Spinal Cord Injury Centre of Western Denmark
Locations (2):
- Denmark (2):
  - Department of Spinal Cord Injuries, Hornbæk
  - Spinal Cord Injury Centre of Western Denmark, Viborg